CLINICAL TRIAL: NCT07303101
Title: One-stage Exchange in Candida Periprosthetic Infection a Suitable Way to go
Acronym: CPCI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9477
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Candida Infection
Keywords: Candida infection; Prosthesis replacement
MeSH Terms: conditions — Candidiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Accounting for only 0.7% to 3% of joint prosthesis infections, yeast infections are considered particularly difficult to treat. They are primarily caused by Candida yeasts, representing over 90% of cases.

Surgical treatment is the cornerstone of managing periprosthetic infections. In cases of chronic bacterial infections, complete implant replacement is necessary and can be performed either in one or two stages.

However, for chronic Candida spp. infections, two-stage prosthesis replacement remains the preferred option. Only three retrospective, single-center studies have evaluated the success rate of one-stage prosthesis replacement in periprosthetic Candida spp. infections in selected patients. Although the sample sizes of these studies are small, the 2-year success rate of 63% to 81% differs little from that of two-stage implant replacement (47% to 100%). Furthermore, systemic antifungal treatment is poorly defined. Recommendations are based on studies with a low level of evidence. The hypothesis is that a single-stage prosthesis replacement combined with appropriate antifungal treatment for chronic periprosthetic Candida spp. infection has the same outcome as a two-stage prosthesis replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years at the time of prosthesis revision
* Operated on at the Strasbourg University Hospitals (HUS) between January 1, 2013, and December 31, 2021
* Hip or knee prosthesis revision
* Possible or proven periprosthetic Candida spp. infection according to the EBJIS diagnostic criteria
* Minimum of 3 deep samples (joint fluid, preoperative sample, and/or prosthesis sonication)

Exclusion Criteria:

* Patient undergoing lavage, synovectomy, and implant preservation
* Patient not receiving systemic antifungal treatment after prosthesis replacement
* Patient with another proven Candida spp. infection or infective endocarditis
* Patient for whom suppressive therapy was prescribed prior to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subject having hip or knee prosthesis revision
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Candida spp. infection eradication rate | for the duration of hospital stay, up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Orthopédique Septique - CHU de Strasbourg - France, Strasbourg, France